CLINICAL TRIAL: NCT02617602
Title: Goal Directed Hemodynamic Management of Acute Heart Failure After Cardiac Surgery in Children: a Prospective Randomised Trial
Brief Title: Goal Directed Hemodynamic Management of Acute Heart Failure After Cardiac Surgery in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDT1.0
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Cardiac Surgery
Keywords: Congenital heart defect; Cardiopulmonary bypass; Goal directed therapy; Acute heart failure
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Goal directed therapy (Experimental): Based on transpulmonary thermodilution, hemodynamic management will be implemented to achieve predefined goals
  Interventions: Procedure: Goal directed therapy
- Control (Active Comparator): Conventional therapy
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Goal directed therapy — Based on transpulmonary thermodilution data, the following interventions will be implemented:
  Global end diastolic volume (GEDV) ≤ 430 ml/m2 and extravascular water index (EVWI) ≤ 10 ml/kg: fluid load; GEDV ≥ 550 ml/m2 and EVWI ≥ 10 ml/kg: furosemide;
  cardiac index (CI) ≤ 2 l/min/m2 - inotropic support:
  * decreased heart rate (HR): dobutamine, dopamine;
  * normal or increased HR: epinephrine, norepinephrine; CI ≥ 2 l/min/m2 and normovolemia: phenylephrine.
  Arms: Goal directed therapy
Other: Control
  Arms: Control

SUMMARY:
Goal directed therapy (GDT) utilises various monitoring techniques to assess cardiovascular performance and allows for timely interventions based on predetermined algorithms. The aim of this prospective randomised study is to evaluate the effect of GDT on major complications in children undergoing radical correction of congenital heart defects, complicated by acute heart failure. Goal directed therapy will be implemented with the aid of transpulmonary thermodilution and based on predetermined algorithms.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent signed by legal representative (parent or guardian)
* radical correction of congenital heart defect(s)
* use of cardiopulmonary bypass
* vasoactive-inotropic Score of 10 or greater during first 24 hours after surgery.

Exclusion Criteria:

* confirmed intranatal infection;
* gestational age < 37 weeks;
* inotropic support prior to surgery;
* acute renal or hepatic failure prior to surgery;
* participation in conflicting randomised controlled studies.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Major complications | Through study completion, an average of 30 days
  Composite of all-cause mortality, extracorporal membrane oxygenation use, cardiac arrest, renal impairment (pRIFLE score of "injury" or higher), sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lomivorotov, PhD, Principal Investigator — Novosibirsk Research Institute of Cirulation Pathology
Locations (1):
- Novosibirsk Research Institute of Circulation Pathology, Novosibirsk, Russia